CLINICAL TRIAL: NCT03616223
Title: A Phase 1/2 Randomized, Double-blind, Placebo-controlled Single Dose Study at Two Dose Levels of FX-322 Administered by Intratympanic Injection in Adults With Stable Sensorineural Hearing Loss
Brief Title: FX-322 in Sensorineural Hearing Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frequency Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX-322-201
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Sensorineural Hearing Loss
Keywords: Intratympanic Administration; Hearing Restoration
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FX-322 Low Dose (Experimental): Cohort of 8. Single intratympanic injection
  Interventions: Drug: FX-322
- FX-322 High Dose (Experimental): Cohort of 8. Single intratympanic injection
  Interventions: Drug: FX-322
- Placebo-Low Dose (Placebo Comparator): Cohort of 4. Single intratympanic injection
  Interventions: Drug: Placebo
- Placebo-High Dose (Placebo Comparator): Cohort of 4. Single intratympanic injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FX-322 — Intratympanic injection of FX-322 consists of laduviglusib and sodium valproate
  Arms: FX-322 High Dose; FX-322 Low Dose
Drug: Placebo — Intratympanic injection
  Arms: Placebo-High Dose; Placebo-Low Dose

SUMMARY:
This is a phase 1/2 study of FX-322 at two dose levels compared to placebo in male and female adults otherwise healthy with stable sensorineural hearing loss.

DETAILED DESCRIPTION:
Sensorineural hearing loss (SNHL) accounts for about 90% of all cases of hearing loss. The study will assess the safety of FX-322 (laduviglusib and sodium valproate) given as a single intratympanic injection in subjects with a medical history of sensorineural hearing loss that is associated with noise exposure or sudden hearing loss. Safety will be evaluated both systemically (lab and clinical monitoring) and locally (otoscopy and audiometry) in 24 subjects, and a blood PK profile of FX-322 will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18-65 years.
2. Established diagnosis of stable sensorineural hearing loss (no changes of 10 dB or more at any frequency) by standard audiometric measures for >6 months.
3. Documented medical history consistent with hearing loss being caused by noise exposure or sudden sensorineural hearing loss (documented audiogram at least 6 months prior to screening required).
4. Female subjects must be of non-childbearing potential or will need to utilize two methods of highly effective contraception during the study participation (e.g. hormonal contraception or an intrauterine device and condoms) or remain abstinent. Male subjects should use condoms with spermicide during the course of the study or remain abstinent. Subjects should not donate sperm or ova during the study period.

Exclusion Criteria:

1. Perforation of tympanic membrane or other tympanic membrane disorders that would interfere with the delivery and safety assessment of an intratympanic medication or reasonably be suspected to affect tympanic membrane healing after injection in either ear. This includes a current tympanostomy tubes.
2. Any conductive hearing loss of 10 dB or more at two or more frequencies in either ear.
3. A pure tone average of 70 dB or greater at 500Hz, 1000Hz, 2000Hz, and 4000Hz in the ear to be injected.
4. Active chronic middle ear disease or a history of major middle ear surgery, as an adult, in the ear to be injected.
5. Subject has had an intratympanic injection in either ear within 6 months of the screening visit.
6. History of clinically significant vestibular symptoms at the discretion of the investigator.
7. History of clinically significant systemic autoimmune disease (e.g. rheumatoid arthritis, Sjogren's syndrome, multiple sclerosis, psoriasis).
8. History of head or neck radiation treatment or exposure.
9. History of substance abuse within 2 years of the Screening Visit.
10. Positive urine pregnancy test or breast-feeding.
11. Any known factor, condition or disease that, in the view of the investigator, might interfere with treatment compliance, study conduct or interpretation of the results such as psychiatric disease or suicidal tendencies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Atiee, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

REFERENCES:
- See also: Journal article — https://journals.lww.com/otology-neurotology/Fulltext/2021/08000/Improved_Speech_Intelligibility_in_Subjects_With.14.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 participants who met all inclusion criteria and no exclusion criteria were enrolled at a single clinic site.
Pre-assignment Details: 23 participants were randomized into one of four treatment groups using a 1:1 allocation ratio for dose cohort (approximately 12 in each cohort) and a 2:1 allocation ratio for study drug (approximately 8 FX-322:4 placebo) within each cohort. Subjects received a single dose of FX-322L (0.05mL), FX-322H (0.2mL), or matching placebo.
Groups:
- Placebo-Low Dose; Placebo-High Dose: Single intratympanic injection of placebo into affected ear
- FX-322 Low Dose: Single intratympanic injection of FX-322 (laduviglusib 0.157mg/sodium valproate 4.43mg) into affected ear
- FX-322 High Dose: Single intratympanic injection of FX-322 (laduviglusib 0.628mg/sodium valproate 17.72mg) into affected ear
Period: Overall Study
Arm/Group | Placebo-Low Dose | Placebo-High Dose | FX-322 Low Dose | FX-322 High Dose
Started | 4 | 4 | 7 | 8
Completed | 4 | 4 | 7 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Low Dose | Placebo-High Dose | FX-322 Low Dose | FX-322 High Dose | Total
Number analyzed (Participants) | 4 | 4 | 7 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 7 | 8 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 9
  Male | 2 | 2 | 5 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 2 | 6
  Not Hispanic or Latino | 3 | 3 | 5 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 6 | 7 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 7 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Event(s) (TEAEs)
Description: Treatment-emergent adverse events (TEAE) were defined as any untoward medical occurrence in a subject administered study drug that does not necessarily have a causal relationship with the treatment and were collected from the time of first dose through end of study (day 90). In particular, audiometric and otoscopic TEAEs were recorded per the American Speech-Language-Hearing Association (ASHA) guidelines.
Time Frame: Baseline through Day 90
Population: Safety Analysis Set = All subjects exposed to study drug and analyzed according to the actual treatment received regardless of the randomized treatment
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo: All participants receiving placebo
Arm/Group | Placebo-Low Dose | Placebo-High Dose | Pooled Placebo | FX-322 Low Dose | FX-322 High Dose
Number analyzed (Participants) | 4 | 4 | 8 | 7 | 8
Participants | 2 | 3 | 5 | 6 | 7

2. Secondary Outcome: Cmax
Description: Maximum concentration (Cmax) of FX-322 (Laduviglusib and Sodium Valproate) directly from individual concentration-time data
Time Frame: Data points taken pre-dose and 0.5, 1, 2, 4, 8, 24 hours post-dose
Population: Pharmacokinetic Analysis Set = All subjects in the Safety Analysis Set with measurable plasma concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FX-322 Low Dose | FX-322 High Dose
Number analyzed (Participants) | 7 | 8
ng/mL
  Cmax of laduviglusib | 0.62 (0.191) | 0.967 (0.361)
  Cmax of sodium valproate | 345 (94.9) | 767 (309)

3. Secondary Outcome: Tmax
Description: Time to reach maximum concentration of FX-322 (Laduviglusib and Sodium Valproate) directly from individual concentration-time data
Time Frame: Data points taken pre-dose and 0.5, 1, 2, 4, 8, 24 hours post-dose
Population: Pharmacokinetic Analysis Set = All subjects in the Safety Analysis Set with measurable plasma concentrations
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | FX-322 Low Dose | FX-322 High Dose
Number analyzed (Participants) | 7 | 8
hr
  Tmax of laduviglusib | 0.95 (0.206) | 1.63 (1.06)
  Tmax of sodium valproate | 2.88 (2.49) | 2.38 (1.06)

4. Secondary Outcome: AUClast
Description: Area under the concentration-time curve of FX-322 (Laduviglusib and Sodium Valproate) from time zero to the time of the last quantifiable concentration, calculated using the linear trapezoidal rule
Time Frame: Data points taken pre-dose and 0.5, 1, 2, 4, 8, 24 hours post-dose
Population: Pharmacokinetic Analysis Set = All subjects in the Safety Analysis Set with measurable plasma concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | FX-322 Low Dose | FX-322 High Dose
Number analyzed (Participants) | 7 | 8
ng*hr/mL
  AUClast of laduviglusib | 1.71 (0.766) | 3.52 (1.31)
  AUClast of sodium valproate | 2730 (2790) | 13100 (4390)

5. Secondary Outcome: t1/2
Description: The observed terminal elimination half-life of FX-322 (Laduviglusib and Sodium Valproate)
Time Frame: Data points taken pre-dose and 0.5, 1, 2, 4, 8, 24 hours post-dose
Population: Pharmacokinetic Analysis Set = Subjects in the Safety Analysis Set with plasma concentrations above the limit of quantification. Concentration-time data below the limit of quantification (BLQ) were treated as zero. The values of 4 of 7 subjects in the low dose group and 2 of 8 subjects in the high dose group were BLQ and were thus excluded from the PAS for t1/2 as those values could not be calculated. The number analyzed for each data point below reflects quantifiable levels within in each group
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | FX-322 Low Dose | FX-322 High Dose
Number analyzed (Participants) | 3 | 6
hr
  t1/2 of laduviglusib: number analyzed (Participants) | 3 | 2
  t1/2 of laduviglusib | 2.58 (0.878) | 2.47 (0.280)
  t1/2 of sodium valproate: number analyzed (Participants) | 2 | 6
  t1/2 of sodium valproate | 14.7 (3.86) | 20.1 (2.93)

6. Secondary Outcome: CL/F
Description: Apparent total body clearance after extravascular administration of FX-322 (Laduviglusib and Sodium Valproate)
Time Frame: Data points taken pre-dose and 0.5, 1, 2, 4, 8, 24 hours post-dose
Population: Pharmacokinetic Analysis Set = Subjects in the Safety Analysis Set with plasma concentrations above the limit of quantification. Concentration-time data below the limit of quantification (BLQ) were treated as zero. The values of 4 of 7 subjects in the low dose group and 2 of 8 subjects in the high dose group were BLQ and were thus excluded from the PAS for CL/F as those values could not be calculated. The number analyzed for each data point below reflects quantifiable levels within in each group
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | FX-322 Low Dose | FX-322 High Dose
Number analyzed (Participants) | 3 | 6
L/hr
  CL/F of laduviglusib: number analyzed (Participants) | 3 | 2
  CL/F of laduviglusib | 54.4 (9.93) | 147 (21.7)
  CL/F of sodium valproate: number analyzed (Participants) | 2 | 6
  CL/F of sodium valproate | 0.510 (0.287) | 0.788 (0.308)

ADVERSE EVENTS:
Time Frame: Baseline through Day 90
Description: Safety Analysis Set = All subjects exposed to study drug and analyzed according to the actual treatment received regardless of the randomized treatment
Arm/Group | Placebo-Low Dose | Placebo-High Dose | Pooled Placebo | FX-322 Low Dose | FX-322 High Dose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4 | 5/8 | 6/7 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Low Dose (N=4) | Placebo-High Dose (N=4) | Pooled Placebo (N=8) | FX-322 Low Dose (N=7) | FX-322 High Dose (N=8)
Ear Discomfort (Ear and labyrinth disorders) | 1 | 1 | 2 | 5 | 4
Ear Pain (Ear and labyrinth disorders) | 1 | 2 | 3 | 1 | 3
Deafness (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 1
Ear Pruritus (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 0
Paraesthesia Ear (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Tympanic Membrace Perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Injection Site Pain (General disorders) | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs must obtain sponsor's written consent before publishing or presenting the trial results.

DOCUMENTS (2):
  • Study Protocol (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT03616223/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03616223/SAP_001.pdf